CLINICAL TRIAL: NCT06893042
Title: A Prospective Study on the Real Word of Acute Liver Failure in Children
Brief Title: Clinical Study of Pediatric Acute Liver Failure
Status: Enrolling by invitation | Type: Observational
Sponsor: Fansen Zeng (Other)
Responsible Party: Sponsor-Investigator, Fansen Zeng, associate chief physician, Guangzhou Women and Children's Medical Center
Organization: Guangzhou Women and Children's Medical Center (Other)
Other Study IDs: 346A01
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-08

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to understand the etiology, prognosis and influencing factors of acute liver failure in children, evaluate the predictive value of children's SOFA score, PELD score and LIU score for the short-term mortality rate of children's liver failure and the infection of children's acute liver failure; analyze the bleeding and kidney damage of children's acute liver failure, and evaluate the quality of life of children's acute liver failure.

DETAILED DESCRIPTION:
PALF is a seriously life-threatening acute disease with a rapid onset, rapid progression and high mortality rate. Especially under the influence of multiple organ dysfunction syndrome (MODS) or other serious complications, clinical prognosis evaluation and treatment decision-making face great challenges.It aims to accurately evaluate the survival probability or liver transplantation needs of patients based on clinical data and biological indicators, and deeply reveal the impact of different factors on the prognosis of PALF from the perspective of etiology, treatment mode (such as mechanical ventilation and plasma replacement) and complications (such as MODS and its score), so as to provide a scientific basis for identifying high-risk groups, optimizing personalized treatment strategies and early diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* （1) The age is less than 18 years old; (2) Acute onset (≤8 weeks), no liver disease basis in the past; (3) Biochemical evidence of severe liver injury ; (4) Coagulation dysfunction that cannot be corrected by vitamin K: prothrombin time (PT) ≥15s or international standardized ratio (INR) ≥1.5, and accompanied by hepatic encephalopathy at the same time; or meet any of PT≥20s, INR≥2.0, may not be accompanied by hepatic encephalopathy; (5) Provide complete clinical data and treatment records. (6) Agree to participate in this study and obtain informed consent.

Exclusion Criteria:(1) Multiple organ failure caused by non-hepatic diseases; (2) Missing data or incomplete follow-up information.

-

Ages: 1 Minute to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The children under the age of 18 diagnosed with acute liver failure in Guangzhou Women's and Children's Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
With the changes of various indicators such as blood ammonia albumin lactic acid coagulation function with the implementation of treatment | From enrollment to the end of treatment at 6 months
  All are specific numerical measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women's and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2026/09/01-2031/09/01